CLINICAL TRIAL: NCT00098631
Title: A Phase II Study Of GW572016 In Squamous Cell Carcinoma Of The Head And Neck (SCCHN)
Brief Title: Lapatinib in Treating Patients With Recurrent and/or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02636; NCI-2012-02636 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000398163; UCCRC-13394; NCI-6718; 13394A (Other: University of Chicago Comprehensive Cancer Center); 6718 (Other: CTEP); N01CM62201 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Lapatinib

ARMS (1):
- Treatment (lapatinib ditosylate) (Experimental): Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth. This phase II trial is studying how well lapatinib works in treating patients with recurrent and/or metastatic head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall response rate in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck treated with lapatinib.

II. Determine the progression-free survival, time to progression, and overall survival of patients treated with this drug.

III. Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 cohorts according to prior epidermal growth factor receptor-targeted therapy (yes vs no).

Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 40-88 patients (21-50 epidermal growth factor receptor [EGFR] inhibitor-naive patients [cohort A] and 19-38 EGFR inhibitor-pre-treated patients [cohort B]) will be accrued for this study within 4-12.6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck

  * Recurrent and/or metastatic disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No more than 2 prior treatment regimens for recurrent or metastatic disease

  * Prior chemotherapy as part of initial curative intent therapy (e.g., neoadjuvant, adjuvant, or concurrent chemotherapy) is allowed and does not count as prior therapy for recurrent or metastatic disease
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance > 60 mL/min
* Cardiac ejection fraction normal by echocardiogram or MUGA
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Able to swallow and retain oral or feeding tube-administered medication
* No malabsorption syndrome
* No requirement for IV alimentation
* No uncontrolled inflammatory gastrointestinal disease (e.g., Crohn's disease or ulcerative colitis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to lapatinib
* No other uncontrolled illness
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* Prior cetuximab allowed
* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior cumulative anthracycline therapy ≥ 450 mg/m^2 of doxorubicin or equivalent
* More than 4 weeks since prior radiotherapy
* No prior surgical procedure affecting absorption
* Recovered from prior therapy
* Other prior epidermal growth factor receptor inhibitors (e.g., gefitinib or erlotinib) allowed
* Concurrent oral anticoagulants (e.g., warfarin) allowed provided there is increased vigilance in monitoring INR
* No concurrent CYP3A4 inhibitors or inducers
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2004-10; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate by RECIST | Up to 6 years
  The 95% confidence intervals should be provided.
Progression-free survival (PFS) | From start of treatment to time of disease progression, assessed up to 6 years
  Will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Overall survival | Up to 6 years
  Will be estimated using the Kaplan-Meier method.
Changes in EGFR, pEGFR, HER2 | Baseline and 12 weeks
  Paired t-tests or Wilcoxon signed rank tests will be performed to examine the magnitude and significance of pre-post treatment changes. To determine whether these markers are correlated with tumor response, both the baseline levels and the pre-post changes will be compared between responders and non-responders using the nonparametric, Wilcoxon rank-sum test. The correlative data will also be entered as covariates into a Cox regression model to determine whether they are predictive of progression-free and overall survival.
Adverse events assessed using NCI CTCAE version 3.0 | Up to 6 years
  Adverse events will be summarized by type and grade.

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States